CLINICAL TRIAL: NCT05262361
Title: Functional Mechanism of Neural Control in Persistent Post-Concussion Symptoms Convergence Insufficiency
Brief Title: Persistent Post-Concussion Symptoms With Convergence Insufficiency
Acronym: PPCS-CI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Jersey Institute of Technology (Other)
Collaborators: Salus University (Other); Children's Hospital of Philadelphia (Other); National Eye Institute (NEI) (NIH); Rutgers University (Other)
Responsible Party: Principal Investigator, Dr. Tara Lynn Alvarez, Professor, New Jersey Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2R01EY023261 (NIH); 2R01EY023261 (NIH)
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Persistent Post-concussive Symptoms; Convergence Insufficiency; Mild Traumatic Brain Injury; Concussion, Mild; Concussion; Eye
MeSH Terms: conditions — Ocular Motility Disorders; Brain Concussion

STUDY DESIGN:
Intervention Model Description: The are two arms. Arm 1 will have participants will have office-based vergence and accommodative therapy (twice per week) immediately after enrollment while arm 2 will have participants have a 6 week delay before enrollment of therapy. There are three assessments: baseline, outcome 1 which is at 6 weeks (arm 1 would be after 12 sessions of therapy and arm 2 would not have participants in vision therapy yet), and outcome 2 which after vision therapy.
Who Masked: Outcomes Assessor
Masking Description: The optometrist will be masked for all outcome assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Office based Vergence and Accommodative Therapy immediately after enrollement (Experimental): This arm will start immediately after baseline assessment. The participant will have two sessions of one hour each for 6 weeks (12 office-based vergence and accommodative therapy sessions). The first outcome measurement will be attained by a masked optometrist. Then, the participant will have 2 more weeks of therapy (4 office-based vergence and accommodative therapy sessions). The second and final outcome measurement will be attained. Assessments include a masked optometric vision exam, objective eye movement recordings and an functional MRI scan.
  Interventions: Behavioral: Office-based Vergence and Accommodative Therapy
- Office based Vergence and Accommodative Therapy Delay 6 weeks post enrollment (No Intervention): This arm will start with a 6 week delay (no vision therapy) after baseline assessment to evaluate natural recovery. After 6 weeks, the first outcome assessment will be attained by a masked optometrist. The participant will have two sessions of one hour each for 8 weeks (16 office-based vergence and accommodative therapy sessions). The second and final outcome measurement will be attained. Assessments include a masked optometric vision exam, objective eye movement recordings and an functional MRI scan.

INTERVENTIONS:
Behavioral: Office-based Vergence and Accommodative Therapy — Office-based Vergence and Accommodative Therapy has four phases which start with gross vergence and accommodation. Disparity vergence is isolated using instruments such as vectograms and accommodation is isolated using near far charts and accommodative rock. The final phase includes the integration of vergence and accommodation to increase range and visual comfort which performing activities close to the person.
  Arms: Office based Vergence and Accommodative Therapy immediately after enrollement

SUMMARY:
Our successful R01 discovered 1) the neural mechanistic difference between typically occurring convergence insufficiency (TYP-CI) and binocularly normal controls and 2) the underlying mechanism of office-based vergence and accommodative therapy (OBVAT) that is effective in remediating symptoms. Adolescent and young adult concussion is considered a substantial health problem in the United States where our team has shown that about half of patients with persistent post-concussion symptoms have convergence insufficiency (PPCS-CI), causing significant negative impact associated with reading or digital screen-related activities, and is believed to be one factor causing delayed recovery impacting return to school, sports, or work. The results of this randomized clinical trial will impact the lives of adolescents and young adults with PPCS-CI to guide professionals on how to manage and treat those with PPCS-CI by 1) comparing the differences between PPCS-CI and TYP-CI, 2) discovering the neural mechanism of OBVAT for PPCS-CI compared to standard-community concussion care, and 3) determining the effectiveness of 12 one-hour sessions compared to 16 one-hour sessions of OBVAT.

DETAILED DESCRIPTION:
During the past 6 years, our study team investigated the neural mechanism of typically-occurring convergence insufficiency (TYP-CI), the most common binocular vision disorder in children and young adults (3.4% to 12.7%5-11). We conducted the only randomized clinical trial (RCT) integrating objective eye movement and fMRI outcome measures, achieving 100% planned enrollment and retention of 100 young adults. Our results localized the reduction in functional activity for TYP-CI compared to controls within the oculomotor vermis (OVM) and the cuneus. Functional activity in the OVM and cuneus was significantly correlated to convergence peak velocity providing the first mechanistic identification of these deficits that create significant burden to those afflicted. Our longitudinal results discovered that the neural mechanistic change stimulated by office-based vergence /accommodative therapy (OBVAT) is an increase in the frontal eye field (FEF) and thalamus functional activity. Increased functional activity from the FEF and thalamus significantly correlates to convergence peak velocity. Results are leading to personalized point-of-care therapies remediating the debilitating symptoms for TYP-CI patients. While our research and results of other RCTs show that OBVAT is the most effective treatment for remediating symptoms and improving vision function in both TYP-CI children and adults, none of these participants had a history of head injury, a pathology that has been linked to CI. Our research team has demonstrated that the prevalence of CI is higher (38% to 49%) in children and adults with persistent post-concussive symptoms (PPCS-CI), than in the non-concussed population. Currently, there is no validated treatment for PPCS-CI. This difference in prevalence, mode of onset (longstanding versus sudden onset), and severity of the condition has led to a debate about whether the diagnostic and management procedures effective for TYP-CI should be utilized for PPCS-CI, and strongly suggests that new research is needed to optimize PPCS-CI management. We are uniquely positioned to provide answers to these questions by building on our work establishing the neurofunctional mechanism of TYP-CI and OBVAT administered to TYP-CI. Such research is of great importance because PPCS-CI is associated with debilitating visual symptoms impacting the return to school/sports, work, or driving. We have identified three significant gaps for the treatment of PPCS-CI that must be addressed to determine its most effective management. First, given the obvious differences in etiology, are there significant differences between TYP-CI and PPCS-CI related to objective eye movement measures (peak velocity, final amplitude, and repeatability) due to underlying neural mechanistic differences? Second, what is the underlying neural mechanism of OBVAT for PPCS-CI compared to TYP-CI? Third, how effective is OBVAT for PPCS-CI and is the dosage of administration different than TYP-CI? This renewal addresses these gaps in clinical science.

ELIGIBILITY:
Inclusion Criteria:

* Between 11 to 35 years
* Concussion diagnosed by a clinical 1 to 6 months ago
* Best-corrected visual acuity of 20/25 in both eyes at distance and near
* willing to wear glasses or contact to correct refractive error if needed
* Global stereopsis of 500 sec of arc or better and 70 sec of arc of better using Randot Stereo Test
* Diagnosis of convergence insufficiency from an optometrist defined as near point of convergence of greater than or equal to 6 cm, positive fusional vergence at 40 cm not meeting Sheard's criteria of at least twice the near phoria or a range of less than or equal to 15 prism diopters, and a convergence insufficiency symptom survey score of 21 or greater for adults or 16 or greater for children.

Exclusion Criteria:

* History of performing office or home-based vision therapy, orthoptics, home-based near target push-ups, or pencil push ups
* Amblyopia (lazy eye) or constant strabismus or strabismus surgery
* Any conditions or diseases that affect accommodation, vergence or ocular motility, such as Multiple Sclerosis, Graves' thyroid disease, Myastheria Gravis, Diabetes, Chemotherapy, or Parkinson's Disease
* Non-removable metal in the body
* Pregnant, planning on becoming pregnant during the study duration, or breastfeeding
* Metal worker

Ages: 11 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-01-19 (Actual); Study Completion 2026-01-19 (Actual)

PRIMARY OUTCOMES:
Near Point of Convergence with Positive Fusional Vergence | after 12 therapy session spanning 6 weeks
  Composite score of how close a participant can view a target a single along midline combined with positive fusional vergence range.

SECONDARY OUTCOMES:
Vergence Peak Velocity | after 12 therapy session spanning 6 weeks
  The maximum speed of a person looking from far to near along midline
Functional Activity within vergence neural circuit | after 12 therapy session spanning 6 weeks
  The amount of blood oxygenation level dependent signal from vergence neural circuit

CONTACTS AND LOCATIONS:
Overall Officials: Tara L Alvarez, PhD, Principal Investigator — New Jersey Institute of Technology
Locations (2):
- United States (2):
  - NJIT, Newark, New Jersey
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
imaging data will be uploaded to FITBIR at the end of the study. Eye movement and clinical data (without any personal identifiers) will be available upon request to the principal investigator (Tara Alvarez, PhD) at the end of the study
Supporting Information: Study Protocol, SAP
Time Frame: after end of study
Access Criteria: FITBIR or email (tara.l.alvarez@njit.edu) to the principal investigator
URL: https://fitbir.nih.gov/

REFERENCES:
- [Derived] Alvarez TL, Scheiman M, Hajebrahimi F, Noble M, Gohel S, Baro R, Bachman JA, Master CL, Goodman A; CONCUSS Investigator Group. CONCUSS randomised clinical trial of vergence/accommodative therapy for concussion-related symptomatic convergence insufficiency. Br J Sports Med. 2025 Oct 1:bjsports-2025-109807. doi: 10.1136/bjsports-2025-109807. Online ahead of print. PMID 41033748
- [Derived] Alvarez TL, Scheiman M, Gohel S, Hajebrahimi F, Noble M, Sangoi A, Yaramothu C, Master CL, Goodman A. Effectiveness of treatment for concussion-related convergence insufficiency: The CONCUSS study protocol for a randomized clinical trial. PLoS One. 2024 Nov 15;19(11):e0314027. doi: 10.1371/journal.pone.0314027. eCollection 2024. PMID 39546477